CLINICAL TRIAL: NCT04833062
Title: The Influence of Advanced Age, Obesity and Diabetes Type on Course and Outcome of Pregnancy With Diabetes Mellitus: Predictive Role of Clinical, Sonographic and Laboratory Findings.
Brief Title: The Influence of Advanced Age, Obesity and Diabetes Type on Course and Outcome of Pregnancy With Diabetes Mellitus.
Status: Not yet recruiting | Type: Observational
Sponsor: Nazarbayev University Medical Center (Other)
Collaborators: City Hospital #2, Nur-Sultan, Kazakhstan (Unknown)
Responsible Party: Sponsor
Organization: Nazarbayev University (Other)
Other Study IDs: 001-2021
Record Dates: First submitted 2021-03-31; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Ultrasonography; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetes mellitus group: Based on DM type, all women will be divided into four groups: prepregnancy/preexisting DM insulin-dependent or independent (types I and II; classes B, C, and D) and gestational DM (GDM) with or without the need for insulin therapy (DM classes A1 and A2). In the case of gestational DM, the gestational week at the time of diagnosis will be registered. We will consider whether women are diagnosed with another preexisting disease (endocrinological or another one) before or during pregnancy, in order to check the relationship of this disease and their DM and potential risks for pregnancy.
  Interventions: Diagnostic Test: Ultrasound; Other: Survey
- Nondiabetic group: Nondiabetic women who received birth assistance at our referral centers and who agreed to participate in the study were included in the control group. A control of healthy (non-diabetic women) mothers so to compare characteristics and outcomes across diabetic groups will comprise the control group.
  Interventions: Diagnostic Test: Ultrasound; Other: Survey

INTERVENTIONS:
Diagnostic Test: Ultrasound — In women presenting for a routine antenatal appointment at 20 gestational weeks an ultrasound assessment will be carried out using the 3.5 MHz abdominal probe in order to assess foetal biometry and anatomy as per the guidelines. We will assess the utility of mid- and third trimester ultrasound parameters for prediction of intrapartal events and perinatal outcomes in patients with diabetes mellitus.
Other: Survey — The maternal baseline characteristics are defined by maternal age at enrollment, parity, number of prenatal visits, some indicators of socioeconomic status and habits, family history of DM (first degree) and prepregnancy hypertension.
  The prepregnancy body mass index (BMI; kg/m2) will be calculated using the self-reported prepregnancy maternal weight; the pregnancy weight gain (kg) will be calculated by the difference between final pregnancy weight and prepregnancy maternal weight and was classified according to the prepregnancy BMI.

SUMMARY:
Results of this project will enable investigators to get information and to compare maternal and pregnancy characteristics and perinatal outcomes of women with different types of Diabetes Mellitus and to identify the independent risk factors for adverse perinatal outcomes. Particularly, the impact of the advanced age, obesity, and type of diabetes on the course and outcome of pregnancy will be evaluated.

DETAILED DESCRIPTION:
The prevalence of obesity and metabolic diseases (such as type 2 diabetes mellitus, dyslipidaemia, and cardiovascular diseases) has increased in recent years, in both industrialized and developing countries. Diabetes mellitus (DM) is one of the most common disorders which occurred during pregnancy. Approximately 15% of pregnancies worldwide are thought to be affected by preexisting or gestational insulin-dependent (type 1) or independent (type 2) diabetes mellitus (DM).

The utility of mid- and third trimester ultrasound parameters will be assessed for prediction of intrapartal events and perinatal outcomes in patients with diabetes mellitus. The importance of mid-trimester uterine artery blood flow and foetal biometry will be investigated for prediction of intrapartal events and perinatal outcomes in patients with diabetes mellitus. Moreover, an investigation of the utility of third trimester (measured at 30 and 34 weeks of gestation) ultrasound scan will be carried out for prediction of intrapartal events and perinatal outcomes in patients with diabetes mellitus. Additionally, researchers will assess the relationship between the cerebro-placental ratio (CPR) and intrapartum and perinatal outcomes in pregnancies complicated by different types of Diabetes mellitus to determine if the CPR measured at 30 and 34 weeks of gestation is predictive of adverse obstetric and perinatal outcomes. At the end, investigators will evaluate the role of the addition of the UAPI to the CPR, alone or as CPUR [cerebro-placental-uterine ratio (CPUR)], in the improvement of the ability of CPR to predict APO at the end of pregnancy in any subgroup of diabetic patients. Finally, this project will enable precise intervention and resource saving as well as provide evidence for preventable targets development.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women with diabetes mellitus (18 yo and older).

Exclusion Criteria:

* Cases of multiple pregnancies
* Cases of long-term use of corticosteroids
* Cases complicated by congenital fetal abnormalities or aneuploidy.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The study will include all pregnant women with diabetes mellitus (DM) that will be followed-up and delivered in our clinics for seven years (from January 1st, 2022 to December 31st, 2028). The data will be prospectively collected and electronically stored at each prenatal visit and each event.
Sampling Method: Non-Probability Sample
Enrollment: 4600 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Mid-trimester ultrasound scan: Foetal biometry | At 20 gestational weeks
  Mid-trimester ultrasound scan will assess foetal biometry [abdominal circumference (AC), femoral length (FL), biparietal dimension (BPD)].
Mid-trimester ultrasound scan: uterine artery blood flow | At 20 gestational weeks
  Mid-trimester ultrasound scan will assess uterine artery blood flow [early-diastolic uterine artery blood flow waveform notching, as well as the uterine artery pulsatility index (UAPI)]
Third trimester ultrasound scan: foetal biometry | At 30 weeks of gestation
  Third trimester ultrasound scan will assess foetal biometry [abdominal circumference (AC), femoral length (FL), biparietal dimension (BPD)].
Third trimester ultrasound scan: foetal biometry | At 34 weeks of gestation
  Third trimester ultrasound scan will assess foetal biometry [abdominal circumference (AC), femoral length (FL), biparietal dimension (BPD)].
Third trimester ultrasound scan: uterine artery blood flow | At 30 weeks of gestation
  The third trimester ultrasound scan will assess uterine artery blood flow [early-diastolic uterine artery blood flow waveform notching, as well as the uterine artery pulsatility index (UAPI)]
Third trimester ultrasound scan: uterine artery blood flow | At 34 weeks of gestation
  The third trimester ultrasound scan will assess uterine artery blood flow [early-diastolic uterine artery blood flow waveform notching, as well as the uterine artery pulsatility index (UAPI)]
Third trimester ultrasound scan: cerebro-placental ratio (CPR) | At 30 weeks of gestation
  This third trimester ultrasound will assess the relationship between the cerebro-placental ratio (CPR) and intrapartum and perinatal outcomes in pregnancies complicated by different types of Diabetes mellitus and to determine if the CPR measured at 30 and 34 weeks of gestation is predictive of adverse obstetric and perinatal outcomes.
Third trimester ultrasound scan: cerebro-placental ratio (CPR) | At 34 weeks of gestation
  This third trimester ultrasound will assess the relationship between the cerebro-placental ratio (CPR) and intrapartum and perinatal outcomes in pregnancies complicated by different types of Diabetes mellitus and to determine if the CPR measured at 30 and 34 weeks of gestation is predictive of adverse obstetric and perinatal outcomes.
Addition of the UAPI to the CPR | At 30 weeks of gestation
  The third trimester ultrasound will assess whether the addition of the UAPI to the CPR, alone or as CPUR [cerebro-placental-uterine ratio (CPUR)], improves the ability of CPR to predict APO at the end of pregnancy in any subgroup of diabetic patients.
Addition of the UAPI to the CPR | At 34 weeks of gestation
  The third trimester ultrasound will assess whether the addition of the UAPI to the CPR, alone or as CPUR [cerebro-placental-uterine ratio (CPUR)], improves the ability of CPR to predict APO at the end of pregnancy in any subgroup of diabetic patients.

CONTACTS AND LOCATIONS:
Overall Officials: Gauri Bapayeva, MD, PhD, Principal Investigator — Nazarbayev University Medical Center

IPD SHARING:
Plan to Share IPD: No